CLINICAL TRIAL: NCT03098589
Title: Revlimid® Capsules Drug Use-results Surveillance Relapsed or Refractory Adult T-cell Leukemia Lymphoma
Brief Title: Revlimid® Capsules Drug Use-results Surveillance (Relapsed or Refractory ATLL)
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-Celgene-JP-PMS-004
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Lymphoma
Keywords: Adult T-cell Leukemia Lymphoma; Teratogenicity; Myelosuppression; Haemorrhage; Infection; Thromboembolism; Hypersensitivity; Tumor lysis syndrome; Peripheral neuropathy; Ischaemic heart disease; Cardiac failure; Arrhythmia; Renal failure; Interstitial lung disease; Hepatic disorder; Hypothyroidism; Gastrointestinal perforation; Orthostatic hypotension; Convulsion; Somnolence; Confusion; Fatigue; Dizziness; Blurred vision; Second primary cancer; Cataract; Revlimid capsules
MeSH Terms: conditions — Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Teratogenesis; Hemorrhage; Infections; Thromboembolism; Hypersensitivity; Tumor Lysis Syndrome; Peripheral Nervous System Diseases; Coronary Artery Disease; Heart Failure; Arrhythmias, Cardiac; Renal Insufficiency; Lung Diseases, Interstitial; Digestive System Diseases; Hypothyroidism; Hypotension, Orthostatic; Seizures; Sleepiness; Confusion; Fatigue; Dizziness; Neoplasms, Second Primary; Cataract | interventions — Lenalidomide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with T-cell leukemia lymphoma treated with Revlimid: Among patients with relapsed or refractory adult T-cell leukemia lymphoma, patients who received Revlimid will be targeted in this surveillance
  Interventions: Drug: Revlimid

INTERVENTIONS:
Drug: Revlimid — Revlimid

SUMMARY:
To understand the safety and efficacy of Revlimid® Capsules 2.5 mg and 5 mg (hereinafter referred to as Revlimid) under actual conditions of use in patients with relapsed or refractory adult T-cell leukemia lymphoma (hereinafter referred to as relapsed or refractory Adult T-cell Leukemia Lymphoma (ATLL)).

1. Planned registration period 3 years
2. Planned surveillance period 4 years and 6 months after a month after the approval for partial changes in the approved items is granted for relapsed or refractory ATLL

ELIGIBILITY:
Inclusion Criteria:

- Relapsed or Refractory Adult T-cell Leukemia Lymphoma

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Among patients with relapsed or refractory adult T-cell leukemia lymphoma (hereinafter referred to as "Adult T-cell Leukemia Lymphoma (ATLL)") who are treated with Revlimid Capsules (hereinafter referred to as "Revlimid", used by both 2.5 mg and 5 mg capsules).
Sampling Method: Probability Sample
Enrollment: 1149 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2020-09-18 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Up to approximately 4 years
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- ASO KK Iizuka Hospital, Iizuka, Fukuoka, Japan